CLINICAL TRIAL: NCT04752189
Title: Preventing Substance Use Among Youth: Behavioral and Economic Impact of Enhanced Implementation Strategies for Communities
Brief Title: Preventing Substance Use Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Andria B Eisman, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-20-10-2821
Record Dates: First submitted 2021-01-23; First posted 2021-02-12 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard MMH Curriculum Implementation (Active Comparator): Teachers will receive the MMH curriculum manual, standard training and as-needed technical assistance, provided to them by the health coordinators; consistent with standard REP.
  Interventions: Behavioral: Standard implementation
- Enhanced Replicating Effective Programs (REP) (Experimental): We will deploy Enhanced REP to include additional tailoring of the MMH curriculum to include trauma-informed approaches, tailored trauma-focused curriculum training, and implementation facilitation, ongoing specialized implementation support.
  Interventions: Behavioral: Enhanced Replicating Effective Programs (Enhanced REP)

INTERVENTIONS:
Behavioral: Enhanced Replicating Effective Programs (Enhanced REP) — Enhanced REP includes 1. a tailored MMH curriculum, 2. tailored training, and 3. ongoing provider consultation or facilitation to support implementation.
  Arms: Enhanced Replicating Effective Programs (REP)
Behavioral: Standard implementation — The standard implementation of the Michigan Model for Health is consistent with Standard REP and includes the curriculum materials, standard training, and as-needed technical assistance.
  Other Names: Standard REP
  Arms: Standard MMH Curriculum Implementation

SUMMARY:
Using a 2-group, mixed method group randomized trial design, this pilot study will compare standard implementation versus Enhanced Replicating Effective Programs (Enhanced REP) to deliver Michigan Model for Health (MMH) in Michigan high schools.

DETAILED DESCRIPTION:
Background: Drug use remains a major public health problem among youth in the United States. Effective implementation of evidence-based interventions for youth is critical for reducing the burden of drug use and its consequences. The Michigan Model for Health (MMH) is an intervention that has demonstrated efficacy in reducing adolescent substance use. Yet, youth rarely receive evidence-based interventions (EBIs) as intended; this is, in part, due to a poor fit between the intervention and the context. The disconnect between the EBI and context is especially pronounced among underserved and vulnerable populations, including among youth exposed to trauma. Trauma is a potent risk factor for substance use, abuse, and the development of substance use disorders. Consequently, we have a critical need to design and test effective, cost-efficient implementation strategies to optimize the fidelity of school-based drug use prevention to better meet the needs of youth exposed to trauma. The objective of this study is to design and test a multi-component implementation strategy to improve intervention-context fit and enhance fidelity and effectiveness.

Methods: Using a 2-group, mixed method, randomized trial design, this pilot study will compare standard implementation (Replicating Effective Programs: REP) versus enhanced Enhanced Replicating Effective Programs (Enhanced REP) to deliver MMH. REP is a previously established implementation strategy that promotes EBI fidelity through a combination of curriculum packaging, training, and as-needed technical assistance. Enhanced REP incorporates tailoring of the EBI package and training and deploys customized implementation support (i.e., implementation facilitation).

This research designs and tests an implementation strategy deployed to systematically enhance the fit between the intervention and the context for a universal drug use prevention curriculum. The proposed research will focus on youth at heightened risk of drug use and its consequences due to trauma exposure. The proposed research is significant because of its potential to have a positive public health impact by preventing and reducing youth drug use and its consequences.

ELIGIBILITY:
Inclusion Criteria:

* Schools which fail to meet state standards for implementation (less than 80% of curriculum) and/or face one or more barriers to MMH implementation

Exclusion Criteria:

* None

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2022-07-14 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Wayne State University, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
From NIH HEAL (Helping to End Addiction Long-term) Public Access and Data Sharing (https://heal.nih.gov/about/public-access-data) information: Electronic copies of publications will be deposited within 4 weeks of acceptance by a journal in PubMed Central with proper metadata to be discoverable and accessible upon publication. Publications will be published under the Creative Commons Attribution 4.0 Generic License (CC BY 4.0) or otherwise dedicated to the public domain. Publications will be made publicly available immediately without an embargo period. Underlying Primary Data for the Publications will be made available through an suitable data repository, such as the NIH HEAL central data repository. To meet program goals, NIH requires broad sharing of Underlying Primary Data from NIH-Supported NIH HEAL Initiative Research Projects in a way that is responsive to concerns about protecting confidential and proprietary data and is consistent with other applicable laws and regulations.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified primary participant (i.e., student) -level data will be available through an appropriate data repository, such as the NIH HEAL Initiative central data repository. The data will be available upon acceptance for publication of the main findings from the final student-level dataset. Data will be available in the NIH HEAL repository per HEAL guidelines.
Access Criteria: Access criteria will be determined by the NIH HEAL guidelines. Access to individual-level data will require entering into a data-sharing agreement that includes requirements to protect participants' privacy and data confidentiality.

REFERENCES:
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] O'neill JM, Clark JK, Jones JA. Promoting mental health and preventing substance abuse and violence in elementary students: a randomized control study of the Michigan Model for Health. J Sch Health. 2011 Jun;81(6):320-30. doi: 10.1111/j.1746-1561.2011.00597.x. PMID 21592127
- [Background] Stirman SW, Miller CJ, Toder K, Calloway A. Development of a framework and coding system for modifications and adaptations of evidence-based interventions. Implement Sci. 2013 Jun 10;8:65. doi: 10.1186/1748-5908-8-65. PMID 23758995
- [Background] Eisman AB, Kilbourne AM, Greene D Jr, Walton M, Cunningham R. The User-Program Interaction: How Teacher Experience Shapes the Relationship Between Intervention Packaging and Fidelity to a State-Adopted Health Curriculum. Prev Sci. 2020 Aug;21(6):820-829. doi: 10.1007/s11121-020-01120-8. PMID 32307625
- [Background] Kilbourne AM, Neumann MS, Pincus HA, Bauer MS, Stall R. Implementing evidence-based interventions in health care: application of the replicating effective programs framework. Implement Sci. 2007 Dec 9;2:42. doi: 10.1186/1748-5908-2-42. PMID 18067681
- [Derived] Eisman AB, Whitman J, Palinkas LA, Fridline J, Harvey C, Kilbourne AM, Hutton DW. A mixed methods partner-focused cost and budget impact analysis to deploy implementation strategies for school-based prevention. Implement Sci Commun. 2023 Nov 9;4(1):133. doi: 10.1186/s43058-023-00511-6. PMID 37946235
- [Derived] Eisman AB, Palinkas LA, Koffkey C, Herrenkohl TI, Abbasi U, Fridline J, Lundahl L, Kilbourne AM. Michigan Model for HealthTM Learning to Enhance and Adapt for Prevention (Mi-LEAP): protocol of a pilot randomized trial comparing Enhanced Replicating Effective Programs versus standard implementation to deliver an evidence-based drug use prevention curriculum. Pilot Feasibility Stud. 2022 Sep 10;8(1):204. doi: 10.1186/s40814-022-01145-6. PMID 36088351
- See also: This website contains the resources for the intervention group and access to the surveys which teachers use to track their lesson fidelity. — http://www.mmhleap.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Schools which failed to meet state standards for implementation (<80% of curriculum) and/or faced one or more barrier to implementation were recruited by Regional School Health Coordinators. Participating teachers taught high school health class.
Pre-assignment Details: 10 schools were assessed for eligibility. 1 school was excluded due to lack of response to eligibility survey and 9 schools were randomized to receive Standard Replicating Effective Programs (REP) or Enhanced REP.
Units Other Than Participants: Schools
Groups:
- Standard REP: Teachers received the digital MMH curriculum, standard training, and as-needed technical assistance, provided to them by the regional school health coordinators.
  Standard implementation: Standard implementation of the Michigan Model for Health is akin to Standard REP and includes the curriculum materials, standard training and as-needed technical assistance.
- Enhanced REP: Teachers in the Enhanced REP group received a tailored MMH curriculum to include trauma-informed approaches, tailored trauma-focused curriculum training, and implementation facilitation (ongoing specialized implementation support).
  Enhanced Replicating Effective Programs (Enhanced REP): Deploy Enhanced REP to optimize the delivery of a drug use prevention intervention in community schools and test its feasibility, acceptability, and appropriateness; Enhanced REP includes tailoring the curriculum, training, and providing ongoing provider consultation, or facilitation, to support implementation.
Period: Overall Study
Arm/Group | Standard REP | Enhanced REP
Started | 369; 5 Schools | 456; 4 Schools
Teacher Participants- Completed Pre-implementation Interview | 5; 5 Schools | 5; 4 Schools
Student Participants- Completed Baseline Student Survey (Students enrolled in the study were a part of the randomized teachers' classrooms.) | 364; 4 Schools | 451; 4 Schools
Teacher Participants - Participated in Interim Interview (Teachers with more than one term of health class in their school participated in an interim interview between semesters. Teachers with only one class per school year were not eligible for an interim interview.) | 1; 1 Schools | 2; 2 Schools
Student Participants- Completed Post-implementation Survey Matched to Baseline Survey (Students were unable to participate in the post-implementation survey if the participating teacher withdrew from the study for any reason.) | 104; 4 Schools | 178; 2 Schools
Teacher Participants- Completed Post-implementation Interview | 4; 4 Schools | 2; 2 Schools
Completed | 108; 4 Schools | 180; 2 Schools
Not Completed | 261; 1 Schools | 276; 2 Schools
Not completed — Withdrawal by Subject | 0 | 150
Not completed — Lost to Follow-up | 261 | 126

BASELINE CHARACTERISTICS:
Units Other Than Participants: Schools
Groups:
- Standard MMH Curriculum Implementation: Standard MMH implementation includes 1. MMH curriculum manual, 2. standard training, and 3. as-needed technical assistance provided by the statewide network of school health coordinators.
  Standard implementation of the Michigan Model for Health is consistent with Standard REP (Replicating Effective Programs)
- Enhanced Replicating Effective Programs (REP): Enhanced REP includes 1. tailored MMH curriculum to include trauma-sensitive content, 2. tailored curriculum training, and 3. implementation facilitation.
  Enhanced Replicating Effective Programs (Enhanced REP): We deploy Enhanced REP to optimize the delivery of a drug use prevention intervention in community schools and test its feasibility, acceptability, and appropriateness.
- Total: Total of all reporting groups
Arm/Group | Standard MMH Curriculum Implementation | Enhanced Replicating Effective Programs (REP) | Total
Number analyzed (Participants) | 369 | 456 | 825
Number analyzed (Schools) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants] — Population: This study includes two separate populations of participants (i.e., teachers and students). We include a separate row for each population group, which adds to the total number of baseline participants
  Participants
    Students: number analyzed (Participants) | 364 | 451 | 815
    Students: <=18 years | 364 | 451 | 815
    Students: Between 18 and 65 years | 0 | 0 | 0
    Students: >=65 years | 0 | 0 | 0
    Teachers: number analyzed (Participants) | 5 | 5 | 10
    Teachers: <=18 years | 0 | 0 | 0
    Teachers: Between 18 and 65 years | 5 | 5 | 10
    Teachers: >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: This study includes two separate populations of participants (i.e., teachers and students). We include a separate row for each population group, which adds to the total number of baseline participants
  Participants
    Man: number analyzed (Participants) | 158 | 226 | 384
    Man: Students | 158 | 226 | 384
    Man: Teachers | 0 | 0 | 0
    Woman: number analyzed (Participants) | 177 | 207 | 384
    Woman: Students | 177 | 207 | 384
    Woman: Teachers | 0 | 0 | 0
    Non-binary: number analyzed (Participants) | 12 | 8 | 20
    Non-binary: Students | 12 | 8 | 20
    Non-binary: Teachers | 0 | 0 | 0
    Other: number analyzed (Participants) | 8 | 6 | 14
    Other: Students | 8 | 6 | 14
    Other: Teachers | 0 | 0 | 0
    Prefer not to say: number analyzed (Participants) | 9 | 4 | 13
    Prefer not to say: Students | 9 | 4 | 13
    Prefer not to say: Teachers | 0 | 0 | 0
    Not collected: number analyzed (Participants) | 5 | 5 | 10
    Not collected: Students | 0 | 0 | 0
    Not collected: Teachers | 5 | 5 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: This study includes two separate populations of participants (i.e., teachers and students). We include a separate row for each population group, which adds to the total number of baseline participants
  Participants
    Black: number analyzed (Participants) | 166 | 211 | 377
    Black: Students | 166 | 211 | 377
    Black: Teachers | 0 | 0 | 0
    White: number analyzed (Participants) | 58 | 100 | 158
    White: Students | 58 | 100 | 158
    White: Teachers | 0 | 0 | 0
    Latino/a: number analyzed (Participants) | 8 | 15 | 23
    Latino/a: Students | 8 | 15 | 23
    Latino/a: Teachers | 0 | 0 | 0
    Native American: number analyzed (Participants) | 6 | 8 | 14
    Native American: Students | 6 | 8 | 14
    Native American: Teachers | 0 | 0 | 0
    Asian American: number analyzed (Participants) | 9 | 9 | 18
    Asian American: Students | 9 | 9 | 18
    Asian American: Teachers | 0 | 0 | 0
    Multiracial: number analyzed (Participants) | 40 | 48 | 88
    Multiracial: Students | 40 | 48 | 88
    Multiracial: Teachers | 0 | 0 | 0
    Unsure: number analyzed (Participants) | 82 | 65 | 147
    Unsure: Students | 77 | 60 | 137
    Unsure: Teachers | 5 | 5 | 10
Region of Enrollment [Number; unit: Schools]
  United States | 5 | 4 | 9
School Size (>1000) [Count of Units; unit: Schools] — Number of schools with more than 1000 students. Population: Publicly available school-level data was used to identify schools with more than 1000 students. Teachers in each school are considered the participants analyzed.
  Schools
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 4 | 3 | 7
Free Reduced Lunch Percentage (>50%) [Count of Units; unit: Schools] — Number of schools where greater than 50% of students receive free and/or reduced lunches. Population: School-level data was used to determine the number of schools in the study which had greater than 50% of students who are eligible to receive free and/or reduced lunches, according to state-level data.
  Schools
    number analyzed (Participants) | 5 | 5 | 10
    (all) | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Indicators of Feasibility
Description: To evaluate comprehensively curriculum feasibility, the investigators used the Consolidated Framework for Implementation Research (CFIR) interview guide to guide the qualitative investigation of using Standard MMH Implementation or MI-LEAP for MMH delivery. The semi-structured interview guide was designed to elicit specific feedback on REP and Enhanced REP components (manual, training, and facilitation) and their feasibility to deliver MMH.
  We used reflexive thematic analysis to generate initial codes guided by the CFIR constructs. To ensure data extracts illustrated the themes and identified the subthemes, we reviewed the themes and subthemes against the original transcripts after the review sessions to ensure the analysis provided a well-organized and thorough view of the data.
  The number of coded interview segments identified during teacher interviews reported here indicate the number of segments from the teacher interviews which align with the identified theme (row title).
Time Frame: 9 months
Population: Teachers who completed the study and participated in interviews. Data collected is from interim- and post-implementation interviews as they pertain directly to the outcome measure.
Measure: Number; unit: Coded interview segments
Units Other Than Participants: Schools
Arm/Group | Standard REP | Enhanced REP
Number analyzed (Participants) | 4 | 2
Number analyzed (Schools) | 4 | 2
Coded interview segments
  Impact of implementation climate on feasibility | 6 | 6
  Impact of strategic implementation leadership on feasibility | 5 | 5

2. Primary Outcome: Indicators of Acceptability
Description: To evaluate comprehensively curriculum acceptability, the investigators used the Consolidated Framework for Implementation Research (CFIR) interview guide to guide the qualitative investigation of using Standard MMH Implementation or MI-LEAP for MMH delivery. The semi-structured interview guide was designed to elicit specific feedback on REP and Enhanced REP components (manual, training, and facilitation) and their feasibility to deliver MMH.
  We used reflexive thematic analysis to generate initial codes guided by the CFIR constructs. To ensure data extracts illustrated the themes and identified the subthemes, we reviewed the themes and subthemes against the original transcripts after the review sessions to ensure the analysis provided a well-organized and thorough view of the data.
  The number of coded interview segments identified during teacher interviews reported here indicate the number of segments from the teacher interviews which align with the identified theme (row title).
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Coded interview segments
Units Other Than Participants: Schools
Groups:
- Standard MMH Curriculum Implementation: Teachers received the digital MMH curriculum, standard training, and as-needed technical assistance, provided to them by the regional school health coordinators.
  Standard implementation: Standard implementation of the Michigan Model for Health is akin to Standard REP and includes the curriculum materials, standard training and as-needed technical assistance.
- Michigan Model for Health: Learning to Enhance and Adapt for Prevention (MI-LEAP): Teachers in the Enhanced REP group received a tailored MMH curriculum to include trauma-informed approaches, tailored trauma-focused curriculum training, and implementation facilitation (ongoing specialized implementation support).
  Enhanced Replicating Effective Programs (Enhanced REP): Deploy Enhanced REP to optimize the delivery of a drug use prevention intervention in community schools and test its feasibility, acceptability, and appropriateness; Enhanced REP includes tailoring the curriculum, training, and providing ongoing provider consultation, or facilitation, to support implementation.
Arm/Group | Standard MMH Curriculum Implementation | Michigan Model for Health: Learning to Enhance and Adapt for Prevention (MI-LEAP)
Number analyzed (Participants) | 5 | 5
Number analyzed (Schools) | 5 | 4
Coded interview segments
  Curriculum materials acceptably met student needs | 46 | 36
  Acceptability of Implementation Facilitation and Support | 6 | 5
  Inner setting influences on curriculum acceptability | 19 | 13

3. Primary Outcome: Indicators of Appropriateness
Description: To evaluate comprehensively curriculum appropriateness, the investigators used the Consolidated Framework for Implementation Research (CFIR) interview guide to guide the qualitative investigation of using Standard MMH Implementation or MI-LEAP for MMH delivery. The semi-structured interview guide was designed to elicit specific feedback on REP and Enhanced REP components (manual, training, and facilitation) and their feasibility to deliver MMH.
  We used reflexive thematic analysis to generate initial codes guided by the CFIR constructs. To ensure data extracts illustrated the themes and identified the subthemes, we reviewed the themes and subthemes against the original transcripts after the review sessions to ensure the analysis provided a well-organized and thorough view of the data.
  The number of coded interview segments identified during teacher interviews reported here indicate the number of segments from the teacher interviews which align with the identified theme (row title).
Time Frame: 9 months
Population: as for outcome 1
Measure: Number; unit: Coded interview segments
Units Other Than Participants: Schools
Arm/Group | Standard MMH Curriculum Implementation | Michigan Model for Health: Learning to Enhance and Adapt for Prevention (MI-LEAP)
Number analyzed (Participants) | 5 | 5
Number analyzed (Schools) | 5 | 4
Coded interview segments
  Appropriateness of curriculum for students | 24 | 29
  Appropriateness of implementation facilitation | 6 | 4

4. Primary Outcome: Incremental Implementation Strategy Cost
Description: We used an activity-based micro-costing approach mapping key activities of Enhanced REP across implementation phases. We used the EPIS (Exploration, Preparation, Implementation, and Sustainment) framework to guide implementation phases and to guide the determination of implementation strategy costs. To accurately assess the time spent on each activity, and therefore the cost, individuals (health coordinators and research staff) recorded time spent on tasks throughout the strategy deployment and documented those activities using an activity log. Because the cost of Enhanced REP is on top of the current practices of Standard REP, we report the incremental cost of Enhanced REP.
Time Frame: 9 months
Measure: Number; unit: Dollars
Units Other Than Participants: Schools
Arm/Group | Enhanced REP | Standard REP
Number analyzed (Participants) | 5 | 4
Number analyzed (Schools) | 4 | 4
Dollars | 11,903 | 0

ADVERSE EVENTS:
Time Frame: 9 Months
Description: AE data was not collected for any group.
Groups:
- Standard MMH Curriculum Implementation: Teachers will receive the MMH curriculum manual, standard training and as-needed technical assistance, provided to them by the health coordinators
  Standard implementation: Standard implementation of the Michigan Model for Health is akin to Standard REP and includes the curriculum materials, standard training and as-needed technical assistance.
- Michigan Model for Health: Learning to Enhance and Adapt for Prevention (MI-LEAP): We will deploy Enhanced REP to include additional tailoring of the MMH curriculum to include trauma-informed approaches, tailored trauma-focused curriculum training, and implementation facilitation, ongoing specialized implementation support.
  Enhanced Replicating Effective Programs (Enhanced REP): Deploy Enhanced REP to optimize the delivery of a drug use prevention intervention in community schools and test its feasibility, acceptability, and appropriateness; Enhanced REP includes tailoring the curriculum, training, and providing ongoing provider consultation, or facilitation, to support implementation.
Arm/Group | Standard MMH Curriculum Implementation | Michigan Model for Health: Learning to Enhance and Adapt for Prevention (MI-LEAP)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT04752189/Prot_SAP_003.pdf
  • Informed Consent Form: Teacher Informed Consent (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04752189/ICF_000.pdf
  • Informed Consent Form: Adolescent Informed Assent (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04752189/ICF_001.pdf
  • Informed Consent Form: Parent Information Letter (2021-08-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT04752189/ICF_002.pdf